CLINICAL TRIAL: NCT03231761
Title: A Randomized Controlled Trial of the Impact of Video Presentations on Medical Students' Explicit and Implicit Attitudes Toward Mental Illness in Nepal
Brief Title: Impact of Video Presentations on Medical Students' Attitudes Toward Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Brandon A Kohrt, MD, PhD, Associate Professor of Psychiatry, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 146/2017
Record Dates: First submitted 2017-07-21; First posted 2017-07-27 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Stigmatization; Depression; Psychosis
MeSH Terms: conditions — Stereotyping; Depression; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Service user testimonial videos (Experimental): Videos with service user testimonials about depression and psychosis
  Interventions: Other: Service user testimonial videos
- mhGAP didactic video (Active Comparator): The intervention in the active comparator arm includes two didactic videos with instruction about depression and psychosis based on the World Health Organization mental health Gap Action Programme (mhGAP) modules for those conditions
  Interventions: Other: mhGAP didactic video
- No video (No Intervention): Participants do not observe any videos prior to the assessment

INTERVENTIONS:
Other: Service user testimonial videos — Service users describe their personal experiences receiving care for depression or psychosis and the impact of the treatment on their quality of life
  Arms: Service user testimonial videos
Other: mhGAP didactic video — Video with a narrated slide presentation describing diagnosis and treatment of depression and psychosis
  Arms: mhGAP didactic video

SUMMARY:
This is a randomized controlled trial examining the impact of videos on medical students' implicit and explicit attitudes and knowledge related to mental illness in Nepal. Medical students are randomized to one of three conditions: (a) no video, (b) a didactic video based on the mental health Gap Action Programme (mhGAP) modules for depression and psychosis; and (c) videos with personal testimonials from mental health service users with depression and psychosis.

DETAILED DESCRIPTION:
Stigma towards mental health patients exists within health systems worldwide, affecting high- and low-income countries alike. Stigmatizing beliefs held by health professionals toward mental illness can have detrimental health impacts on the patients. These stigmatizing beliefs against mental health patients within the health system have been noted across South Asia, including Nepal. Two sources of stigmatizing beliefs towards mental illness are explicit (conscious) and implicit (unconscious) attitudes held by health professionals. There is a dearth of research that investigates both explicit and implicit attitudes of health professionals towards mental health in South Asia though. One method to reduce stigma is through contact with people who suffer from mental illness. However, there is a gap in the literature on low- and middle-income countries integrating contact with mental health service users in health provider trainings. Forthcoming research in Nepal is exploring the causal impact of service user involved mental health trainings of health professionals on explicit and implicit attitudes as well as clinical care, but this research has yet to investigate the effects of service user training on health professional students (in progress). Research efforts on mental health trainings should be expanded to student populations to reduce negative attitudes before providers enter the workforce.

The purpose of this study is to evaluate whether information-based training with or without service user testimony is more effective at reducing implicit and explicit biases toward mental health patients and increasing clinical care in Nepali health professional students. The findings from this study will fill the gap in research that evaluates intervention efficacy of reducing stigma towards mental health patients in Nepali student health education. By implementing mental health trainings, the long-term goals of this intervention are to reduce stigma held by health professionals against mental health patients and improve clinical care in Nepal by reducing negative implicit and explicit attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Medical students in universities in Nepal

Exclusion Criteria:

* Medical students are excluded if they have already completed their psychiatric clinical rotation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Social Distance Scale | Immediately after presentation of experimental, active comparator, or no intervention condition (duration of experimental and active comparator conditions is 15-20 minutes)
  Likert rating scale with items referring to level of social distance from persons with mental illness

SECONDARY OUTCOMES:
Implicit Association Test (IAT) | Immediately after presentation of experimental, active comparator, or no intervention condition (duration of experimental and active comparator conditions is 15-20 minutes)
  Implicit Association Test for biases associating mental illness and physical illness by two attributes: violence and burdensomeness
Modified Community Informant Detection Tool (CIDT) vignettes for diagnostic and treatment knowledge assessment | Immediately after presentation of experimental, active comparator, or no intervention condition (duration of experimental and active comparator conditions is 15-20 minutes)
  Vignettes followed by knowledge assessment (multiple choice and free response questions) to evaluate ability to correctly diagnose and recommend treatment for person with depression and psychosis, based on vignettes from CIDT used in Nepal

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Kohrt, MD, PhD, Principal Investigator — George Washington University
Locations (2):
- Nepal (2):
  - Tribhuvan University Institute of Medicine, Maharajgunj, Kathmandu
  - Kathmandu University School of Medicine, Dhulikhel

IPD SHARING:
Plan to Share IPD: Undecided
Upon request, the researchers will share medical student response data if approved by the principal investigator, and medical school research officials.

REFERENCES:
- [Derived] Tergesen CL, Gurung D, Dhungana S, Risal A, Basel P, Tamrakar D, Amatya A, Park LP, Kohrt BA. Impact of Service User Video Presentations on Explicit and Implicit Stigma toward Mental Illness among Medical Students in Nepal: A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Feb 22;18(4):2143. doi: 10.3390/ijerph18042143. PMID 33671743